CLINICAL TRIAL: NCT07332598
Title: Mayo Clinic Precure - Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Executive Director, Center for Individualized Medicine, Mayo Clinic
Other Study IDs: 25-005869
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Genetic Predisposition; Exposure, Environmental
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Saliva, stool, urine, blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected Genetic Predisposition or Multi-Omics Contribution: Patients with a diagnosis or phenotype with the potential for association with a genetic predisposition or Multi-Omics Contribution
- Health Control: Patients with no diagnosis associated with a genetic predisposition or Multi-Omics Contribution.

SUMMARY:
The goal of this observational study is to 1) better understand and predict biological processes before disease begins or is identified, 2) study genomic and environmental contributors to disease, 3) identify ways to stop disease advancement before it becomes serious or complex, and 4) identify potential targets for disease therapy.

Participants will be asked to:

* collect biological samples,
* download a mobile app,
* collect speech (voice) recordings, and
* complete surveys

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Registered Mayo Clinic patient
* Able to provide informed written consent
* Able to receive mail and packages within a United States (US) state
* Able to collect and ship samples within a US state via FedEx for overnight delivery

Exclusion Criteria:

* Active hematological cancer or history of a hematological cancer
* Allogeneic Bone Marrow Transplant (autologous bone marrow transplant recipients are acceptable if collected at least one month after transplant)
* Other co-morbidity that, in physician's opinion, would interfere with patient's ability to participate in the study (e.g., reduced ability to comprehend, i.e., dementia, intellectual disability, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Build a comprehensive, multi-omics and phenotype dataset | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N. Lazaridis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas DC. High-volume "-omics" technologies and the future of molecular epidemiology. Epidemiology. 2006 Sep;17(5):490-1. doi: 10.1097/01.ede.0000229950.29674.68. No abstract available. PMID 16906051
- [Background] Ramos RG, Olden K. Gene-environment interactions in the development of complex disease phenotypes. Int J Environ Res Public Health. 2008 Mar;5(1):4-11. doi: 10.3390/ijerph5010004. PMID 18441400
- [Background] Wild CP. Complementing the genome with an "exposome": the outstanding challenge of environmental exposure measurement in molecular epidemiology. Cancer Epidemiol Biomarkers Prev. 2005 Aug;14(8):1847-50. doi: 10.1158/1055-9965.EPI-05-0456. No abstract available. PMID 16103423